CLINICAL TRIAL: NCT05253495
Title: Reducing the Burden of Oncologic Chemoradiotherapy And Radiation Exposure From Diagnostic Imaging by Utilizing Targeted Immunotherapy in Children, Adolescents and Young Adults With Lymphoma
Brief Title: Chemoradiotherapy With Targeted Immunotherapy in Pediatric Lymphoma
Acronym: RADICAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14601
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Non-hodgkin Lymphoma; Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1a (Experimental): Mature B-cell Non-hodgkin Lymphoma [MB NHL], GROUP B will receive reduction therapy with dexamethasone, vincristine and cyclophosphamide (DOC), then undergo disease assessment. If tumor reduction ≥ 20%, will get induction 1 and 2 with polatuzumab vedotin, cyclophosphamide, vincristine, methotrexate, rituximab, doxorubicin (Pv-COM3RA25D) 1 and 2, then Consolidation 1 with rituximab, cytarabine, methotrexate (R-CYM) . Patients will undergo disease assessment post Consolidation 1. If no residual disease, they proceed to receive Consolidation 2 with Pv-R-CYM (R-CYM 2).
  Cohort Ia patients with < 20% tumor reduction post DOC will be assigned to Cohort Ib starting at Induction 1. Cohort Ia patients with residual disease post Consolidation 1 will be assigned to Cohort Ib starting at Consolidation 1 polatuzumab vedotin, rituximab, high dose cytarabine, cytarabine, high dose methotrexate, etoposide (Pv-R-CYVE 1).
  Interventions: Drug: DOC Group B; Drug: Pv-COMRAD 1 and 2 Group B; Drug: Pv-R-CYM 1 and 2 Group B
- Cohort 1b (Experimental): MB NHL, GROUP C will receive reduction therapy with DOC. Patients with < 20% tumor reduction will be off protocol. Patients with ≥ 20% tumor reduction get Induction 1 and 2 with cyclophosphamide, doxorubicin, dexamethasone, high dose methotrexate, polatuzumab vedotin, and triple intrathecal chemotherapy (M8A30D CPR) 1 and 2, then Consolidation 1 with Pv-R-CYVE 1. If no residual disease, they get Consolidation 2 (Pv-R-CYVE 2), followed by Maintenance (M) 1 with M8A30D CP, M 2 with Pv-cytarabine/etoposide, M 3 with cyclophosphamide, doxorubicin, dexamethasone and polatuzumab vedotin (A30D CP), and M 4 with Pv-cytarabine/etoposide. Cohort Ib patients with CNS disease will receive additional intrathecal chemotherapy and high dose methotrexate during Consolidation.
  Interventions: Drug: DOC Group C; Drug: MAD CPR 1 and 2; Drug: Pv-R CYVE 1 and 2; Drug: Pv-R CYVE-MTX 1 and 2; Drug: MAD CP; Drug: Pv-Cytarabine/etoposide; Drug: AD CP; Radiation: Involved Site Radiation Therapy
- Cohort 2a (Experimental): Classical Hodgkin lymphoma, INTERMEDIATE RISK will receive 2 cycles of brentuximab vedotin (Bv), doxorubicin, vinblastine, dactinomycin, and rituximab (Bv-AVD-R 1 and 2). Response assessment with FDG-PET scan after 2 cycles of Bv-AVD-R. Rapid early responders (RER) will continue therapy with 2 cycles of Bv, vinblastine, dactinomycin, nivolumab, and rituximab (Bv-NVD-R 1 and 2). RERs will not receive radiation therapy. Patients deemed to be Slow Early Responders (SER) after 2 cycles of Bv-AVD-R will continue therapy with 4 cycles of Bv-NVD-R (Bv-NVD-R 1, 2, 3, and 4). Radiation therapy will be given at completion of therapy only for SER patients NOT achieving complete remission at the end of chemoimmunotherapy.
  Interventions: Drug: Bv-AVD-R 1 and 2: COHORT IIa; Drug: Bv-NVD-R, Cycle 1-2; Drug: Bv-NVD-R, Cycle 1-4 SER
- Cohort 2b (Experimental): COHORT IIb (Classical Hodgkin lymphoma, HIGH RISK) Cohort IIb patients will receive 2 cycles of brentuximab vedotin (Bv), doxorubicin, vinblastine, dactinomycin, and rituximab (Bv-AVD-R 1 and 2). Response assessment will be performed with FDG-PET scan after 2 cycles of Bv-AVD-R. Rapid early responders (RER) will continue therapy with 4 cycles of Bv, vinblastine, dactinomycin, nivolumab, and rituximab (Bv-NVD-R 1, 2, 3, and 4). RERs will not receive radiation therapy. Patients deemed to be Slow Early Responders (SER) after 2 cycles of Bv-AVD-R will receive 2 cycles of Bv, nivolumab, doxorubicin, vinblastine, dactinomycin, and rituximab (Bv-NAVD-R 1 and 2), followed by 4 cycles of Bv, vinblastine, dactinomycin, nivolumab, and rituximab (Bv-NVD-R 1, 2, 3, and 4). Radiation therapy will be given at completion of therapy only for SER patients NOT achieving complete remission at the end of chemoimmunotherapy.
  Interventions: Drug: Bv-AVD-R; Drug: Bv-NVD-R, Cycle 1-4 RER; Drug: Bv-NAVD-R, Cycle 1-2; Radiation: Involved Site Radiation Therapy

INTERVENTIONS:
Drug: DOC Group B — Cyclophosphamide 300 mg x1; dexamethasone x 7; vincristine x1
  Other Names: Reduction Phase
  Arms: Cohort 1a
Drug: Pv-COMRAD 1 and 2 Group B — polatuzumab vedotin x1; dexamethasone x 5; vincristine x1, cyclophosphamide x 3; doxorubicin x1; methotrexate x; rituximab 2x; ITT x1
  Other Names: Induction 1 and 2
  Arms: Cohort 1a
Drug: Pv-R-CYM 1 and 2 Group B — polatuzumab vedotin x 1; methotrexate x 1; rituximab x 1; cytarabine x 5;
  Other Names: Consolidation 1 and 2
  Arms: Cohort 1a
Drug: DOC Group C — cyclophosphamide x 1, dexamethasone x 5; vincristine x1; IT triples x 3
  Other Names: Reduction with IT
  Arms: Cohort 1b
Drug: MAD CPR 1 and 2 — methotrexate x 1; dexamethasone x 5; polatuzumab Vedotin x 1, cyclophosphamide x 3; doxorubicin x 1; rituximab x2; IT triples x 2 in induction 1, IT triples x 2 in induction 2
  Other Names: Induction 1 and 2 Group C
  Arms: Cohort 1b
Drug: Pv-R CYVE 1 and 2 — Polatuzumab Vedotin x 1; Rituximab x 1; Cytarabine x 5; Etoposide x4;
  Other Names: Consolidation 1 and 2 Group C CNS Negative
  Arms: Cohort 1b
Drug: Pv-R CYVE-MTX 1 and 2 — Polatuzumab Vedotin x 1; Rituximab x 1; Cytarabine x 5; Etoposide x4; high dose cytarabine x4; high dose methotrexate x 1 (only consolidation 1); IT triples x 2 (only 1 in consolidation 2)
  Other Names: Consolidation 1 and 2 Group C CNS Positive
  Arms: Cohort 1b
Drug: MAD CP — dexamethasone x1; polatuzumab vedotin x 1; cyclophosphamide x 2; doxorubicin x 1; high dose methotrexate x 1; IT triples x 1
  Other Names: Maintenance 1 Group C
  Arms: Cohort 1b
Drug: Pv-Cytarabine/etoposide — polatuzumab vedotin x 1; cytarabine x 5; etoposide x 3;
  Other Names: Maintenance 2, 4 Group C
  Arms: Cohort 1b
Drug: AD CP — polatuzumab vedotin x 1; cyclophosphamide x2; doxorubicin x 2;
  Other Names: Maintenance 3 Group C
  Arms: Cohort 1b
Drug: Bv-AVD-R 1 and 2: COHORT IIa — brentuximab vedotin x 2; doxorubicin x 2; vinblastine x 2; dacarbazine 2x; rituximab x 2
  Other Names: Intermediate Risk cohort IIa
  Arms: Cohort 2a
Drug: Bv-NVD-R, Cycle 1-2 — brentuximab vedotin x 2; nivolumab x 2; vinblastine x2; dacarbazine x 2; rituximab x 2;
  Other Names: Cohort IIa Rapid Early Responders
  Arms: Cohort 2a
Drug: Bv-NVD-R, Cycle 1-4 SER — brentuximab vedotin x 2; nivolumab x 2; vinblastine x 2; rituximab x 2;
  Other Names: Cohort IIa Slow Early Responders
  Arms: Cohort 2a
Drug: Bv-AVD-R — Brentuximab vedotin x2; doxorubicin x2; vinblastine x 2; dacarbazine x 2; rituximab x2;
  Other Names: High-Risk cohort IIb
  Arms: Cohort 2b
Drug: Bv-NVD-R, Cycle 1-4 RER — brentuximab vedotin x 2; nivolumab x 2; vinblastine x 2; dacarbazine x 2; rituximab x 2;
  Other Names: cohort IIb Rapid Early Responders
  Arms: Cohort 2b
Drug: Bv-NAVD-R, Cycle 1-2 — brentuximab vedotin x 2; nivolumab x 2; doxorubicin x 2; vinblastine x 2; dacarbazine x 2; rituximab x 2;
  Other Names: cohort IIb Slow Early Responders
  Arms: Cohort 2b
Radiation: Involved Site Radiation Therapy — 21 Gy in 14 fractions of 1.50 Gy per day. The treatment will be given 5 days per week. All fields shall be treated once each day. The total elapsed treatment time will be 2.8 weeks (14 sessions) for each field.
  Other Names: Cohort II ONLY
  Arms: Cohort 1b; Cohort 2b

SUMMARY:
The addition of targeted immunotherapy will be safe and well tolerated and facilitate the reduction of anthracycline exposure while preserving lymphoma disease control in children, adolescents and young adults (CAYA) with mature B-cell non-Hodgkin lymphoma (MB-NHL) and classical Hodgkin lymphoma (cHL).

DETAILED DESCRIPTION:
The primary objective is 1) to determine feasibility and safety, as defined by dose limiting toxicities (DLTs), of adding polatuzumab vedotin (Pv) in combination with rituximab (RTX) containing French-American-British (FAB) chemoimmunotherapy, with reduced dose anthracycline, in CAYA with intermediate and high risk newly diagnosed MB-NHL; 2) To define the feasibility and safety, as defined by DLTs, of the addition of nivolumab to the backbone of reduced toxicity chemoimmunotherapy with brentuximab vedotin (Bv), vinblastine, dacarbazine and rituximab, with reduced dose anthracycline, in CAYA with newly diagnosed intermediate and high risk cHL.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with histologically or cytologically proven newly diagnosed MB-NHL or cHL according to WHO Classification who meet the following criteria are eligible:

COHORT I:

Burkitt lymphoma (ICD-O 9687/3) Burkitt-like lymphoma with 11q aberration (ICD-O 9687/3) Diffuse large B-cell lymphoma, NOS (ICD-O 9680/3) High grade B-cell lymphoma (ICD-O 9680/3)

COHORT Ia: stage III with LDH ≥ 2 ULN OR stage IV (5-24% bone marrow lymphoma infiltration) (GROUP B)61

COHORT Ib: any CNS involvement and/or BM involvement (≥ 25% lymphoma cells) (GROUP C)61 OR patients with less than 20% tumor size reduction post chemotherapy with cyclophosphamide, dexamethasone, vincristine (DOC Reduction for Cohort Ia).

COHORT II Classical Hodgkin lymphoma (ICD-O 9650/3, 9663/3, 9651/3, 9652/3, 9653/3)

COHORT IIa: stage I-IIA with bulky ± E, I-IIB no bulky ± E, IIIA ± E (INTERMEDIATE RISK)

COHORT IIb: stage IIB with bulky ± E, IIIA with bulky ± E, IIIB, IV (HIGH RISK)

* Adequate organ function

Exclusion Criteria:

* Primary mediastinal B-cell lymphoma (PMBL)
* T-cell/histiocyte-rich large B-cell lymphoma
* Gray zone lymphoma
* Follicular lymphoma
* Nodular lymphocyte-predominant Hodgkin lymphoma (NLPHL)
* Posttransplant lymphoproliferative lymphoma (PTLD)

Ages: 3 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Grade 3 and 4 Adverse Events related to polatuzumab vedotin | 1 year
  to evaluate the DLTs of polatuzumab vedotin (Pv) in combination with rituximab (RTX) containing French-American-British (FAB) chemoimmunotherapy, with reduced dose anthracycline to MB-NHL
Grade 3 and 4 Adverse events related to nivolumab | 1 year
  To evaluate the DLTs of nivolumab to the backbone of reduced toxicity chemoimmunotherapy with brentuximab vedotin (Bv), vinblastine, dacarbazine and rituximab, with reduced dose anthracycline in intermediate and high risk cHL

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Principal Investigator — New York Medical Center
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - University of Flordia, Gainsville, Florida
  - New York Medical College, Vallhala, New York

IPD SHARING:
Plan to Share IPD: No